CLINICAL TRIAL: NCT06840613
Title: Comparison of Glucophage Plus Myo-Inositol Versus Glucophage in Terms of Glycemic Control Among Patients With Gestational Diabetes Mellitus
Brief Title: Glucophage Plus Myo-Inositol vs Glucophage in Glycemic Control Among Patients With Gestational Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Hifza Rasheed, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp129
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: GDM; Diabetes Mellitus; Pregnancy; Glycemic Control
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Inositol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucophage Plus Myo-Inositol (Active Comparator): Intervention: Patients in this group will receive 2 capsules of Myo-Inositol (2000 mg each) along with 500 mg Glucophage three times a day.
  Monitoring: Blood glucose levels will be measured at baseline and after treatment.
  Interventions: Other: Myo-Inositol; Other: Glucophage
- Glucophage Alone (Active Comparator): Intervention: Patients in this group will receive 500 mg Glucophage three times a day.
  Monitoring: Blood glucose levels will be measured at baseline and after treatment.
  Interventions: Other: Glucophage

INTERVENTIONS:
Other: Myo-Inositol — Intervention: Patients in this group will receive 2 capsules of Myo-Inositol (2000 mg each) along with 500 mg Glucophage three times a day.
  Monitoring: Blood glucose levels will be measured at baseline and after treatment
  Arms: Glucophage Plus Myo-Inositol
Other: Glucophage — Intervention: Patients in this group will receive 500 mg Glucophage three times a day.
  Monitoring: Blood glucose levels will be measured at baseline and after treatment.

SUMMARY:
This randomized controlled trial aims to compare the efficacy of Glucophage plus Myo-Inositol versus Glucophage alone in glycemic control among patients with gestational diabetes mellitus (GDM). The study will assess whether the addition of Myo-Inositol improves glycemic control and reduces insulin requirements in GDM patients. Participants will be randomized into two groups: one receiving Myo-Inositol in combination with Glucophage and the other receiving Glucophage alone. The primary outcome will be glycemic control as assessed by fasting and postprandial glucose levels. Secondary outcomes include insulin requirement and gestational age at initiation of insulin therapy.

DETAILED DESCRIPTION:
This prospective, single-center, randomized controlled trial is designed to evaluate the efficacy of Myo-Inositol supplementation in combination with Glucophage compared to Glucophage alone for glycemic control in women diagnosed with gestational diabetes mellitus (GDM). The trial will be conducted at SIMS/Services Hospital Lahore under the supervision of the University of Health Sciences Lahore.

Gestational diabetes mellitus (GDM) is a condition characterized by glucose intolerance that is first recognized during pregnancy, posing significant health risks for both the mother and fetus. Despite various treatment approaches, achieving optimal glycemic control remains a challenge. While Glucophage (Metformin) is widely used for managing GDM, Myo-Inositol has gained attention for its potential role in improving insulin sensitivity and reducing the need for additional pharmacological interventions.

Study Design and Methodology:

This study will enroll 90 participants aged 18-35 years with singleton pregnancies diagnosed with GDM between 22-32 weeks of gestation.

Participants will be randomly assigned to one of two intervention groups:

Experimental Group (Group A): Patients will receive 2000 mg Myo-Inositol (two capsules) with 500 mg Glucophage, three times a day.

Control Group (Group B): Patients will receive 500 mg Glucophage, three times a day.

All participants will be educated on lifestyle modifications and dietary control, and their blood glucose levels will be monitored throughout the study.

Data will be collected at baseline and at multiple time points during pregnancy to assess glycemic control, the need for insulin therapy, and any adverse effects associated with the interventions.

Rationale for the Study:

Myo-Inositol is an insulin-sensitizing agent that plays a crucial role in glucose metabolism. Emerging evidence suggests that Myo-Inositol supplementation may reduce insulin resistance, lower blood glucose levels, and decrease the likelihood of requiring insulin therapy. By comparing its effects in combination with Glucophage, this study aims to determine whether Myo-Inositol can serve as an effective adjunct therapy for managing GDM.

Expected Outcomes and Implications:

Primary Outcome: Improved glycemic control as measured by fasting and postprandial blood glucose levels.

Secondary Outcomes: Reduction in the number of patients requiring insulin therapy, delayed initiation of insulin if needed, and improved maternal and fetal outcomes.

The results of this study could help shape future clinical guidelines for GDM management, offering a non-invasive, cost-effective alternative to conventional treatment approaches.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 to 35 years and Singleton pregnancy
* GDM diagnosed during pregnancy as per operational definition
* 22 to 32 weeks of gestation
* No more than 35 days after GDM diagnosis
* BMI of 18 to 29
* Capacity for self-monitoring of blood glucose

EXCLUSION CRITERIA:

* Patients with obesity BMI more than or equal to 30.
* Already taking insulin during this pregnancy or oral hypoglycemic agents
* Patients taking long time corticosteroid treatment
* Patients with history of pre-existing diabetes
* Overt diabetes diagnosed during pregnancy, i.e. fasting plasma glucose ≥ 126 mg/dL (7 mmol/l) and/or 2-hour post OGTT plasma glucose value ≥ 200 mg/dL (11.1 mmol)
* History of any bariatric surgery
* Twin pregnanc

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | Baseline and up to 12 weeks
  Glycemic control is defined as fasting glucose <95 mg/dL and postprandial glucose <120 mg/dL.
  Blood glucose levels will be recorded at follow-up visit

IPD SHARING:
Plan to Share IPD: Undecided